CLINICAL TRIAL: NCT06992765
Title: Evaluation of Heysong Japanese Green Tea for Improving Blood Lipid Function
Brief Title: Evaluation of Green Tea for Improving Blood Lipid Profile
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Eagletek Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: lin5611_2
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hypercholesterolemia
Keywords: Green tea; Cholesterol; Triglyceride; Blood lipid
MeSH Terms: conditions — Hypercholesterolemia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 2 bottles of light green tea daily containing totally 108 mg of catechin
  Interventions: Dietary Supplement: Placebo
- Intervention (Experimental): 2 bottles of light green tea daily containing totally 684 mg of catechin
  Interventions: Dietary Supplement: Intervention

INTERVENTIONS:
Dietary Supplement: Intervention — 2 bottles of light green tea daily containing totally 684 mg of catechin
  Arms: Intervention
Dietary Supplement: Placebo — 2 bottles of light green tea daily containing totally 108 mg of catechin
  Arms: Placebo

SUMMARY:
The objects of this study are to evaluate the effects of the "Heysong japanese green tea" on the human subjects who are dyslipidemia. In this trial, 40 healthy subjects whose ages are 18~65 years old (20 for placebo and 20 for experimental) will be included. The total experiment will be 16 weeks and the intervention period will be 12 weeks, within which, at wk 0, 2, 8, 14 and 16, serum triglyceride (TG), total cholesterol (TC), high density lipoprotein cholesterol (HDL-C) and low density lipoprotein cholesterol (LDL-C) values would be measured. Urine/feces samples and anthropometric data will also be acquired. The results will be analyzed according to the methods published by the Ministry of Health and Welfare of Taiwan Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Male and female. Age between 18-65 years old.
* Those who have been assessed as dyslipidemia by a family physician but have not yet required medication. The following measurement values were used as evaluation criteria:

  1. Hypercholesterolemia: plasma total cholesterol (TC) >200 mg/dL;
  2. Mixed hyperlipidemia: plasma total cholesterol (TC) >200 mg/dL , triglyceride (TG) >200 mg/dL;
  3. Hypertriglyceridemia: plasma triglyceride (TG) >200 mg/dL, and high-density lipoprotein cholesterol (HDL-C) < 35 mg/dL or TC/HDL-C >5.

Exclusion Criteria:

* Pregnant, breastfeeding, menopausal women.
* Take any drugs or supplements that can affect blood lipid levels 2 weeks before or during the experiment.
* People with intolerance to caffeine or green tea.
* People who take drugs for chronic diseases.
* People who smoke or drink alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Serum total cholesterol | Wk(-2), Week(0) (Baseline), Wk(6), Wk(12) and Wk(14)
  Total cholesterol is measured by the Department of Laboratory Medicine of Taipei Medical University Hospital (TMUH)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Total cholesterol in serum
Supporting Information: Study Protocol